CLINICAL TRIAL: NCT05245695
Title: Deep Neural Network Stratification for the Use in Detecting Endometriosis in Women Affected by Chronic Pelvic Pain (EndoCheck)
Brief Title: Deep Neural Network Stratification for Use Detecting Endometriosis in Women Affected by Chronic Pelvic Pain (EndoCheck)
Status: Recruiting | Type: Observational
Sponsor: Aspira Women's Health (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-2021
Record Dates: First submitted 2022-02-01; First posted 2022-02-18 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Endometriosis
Keywords: Endometriosis; Biomarkers; Deep neural network
MeSH Terms: conditions — Endometriosis | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Cell-free DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Observational study, no intervention — Observational study, no intervention

SUMMARY:
The goal of this observational study is to determine the clinical validity of a deep neural network algorithm that utilizes protein biomarker detection of Endometriosis - "EndoCheck" - as an "aid in diagnosis" for endometriosis and to show validity as a diagnostic test

DETAILED DESCRIPTION:
The objective is to confirm the clinical performance (sensitivity and specificity) of EndoCheck when compared to laparoscopic surgical assessment as an "aid in diagnosis" for endometriosis in subjects who present with chronic pelvic pain.

The primary endpoint of the study is to optimize the test to achieve the success criteria of at least 94% and 79% sensitivity and specificity, respectively. Secondary endpoints include examining the performance of the test in patients stratified by pain severity and other clinical factors.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to provide written informed consent.
* Participant is a female aged 14 to 50 years old at time of consent.
* Participant is scheduled to undergo laparotomy or laparoscopy for symptomology consistent with possible endometriosis

Exclusion Criteria:

* Participant is a female in a pre-menarchal state.
* Participant is pregnant.
* Participant has an active malignancy.
* Participant is known to have tested positive for human immunodeficiency virus or hepatitis A, B, or C.
* Participant has an active pelvic infection or other infections contraindicated for surgery.
* Participant has participated (±3 months of study enrollment) in a clinical trial where an investigational drug/ device/ procedure was or is planned to be administered.
* Participant has any general health or behavioral condition that, in the opinion of the investigator, should exclude the participant from participation.
* Participant is under 14 years old or over 50 years old

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Women scheduled for a gynecologic surgery
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity | 24 months
  The primary endpoint of the study is to optimize the test to achieve the success criteria of at least 94% and 79% sensitivity and specificity, respectively

SECONDARY OUTCOMES:
Performance | 24 months
  Examining the performance of the test in patients stratified by pain severity and other clinical factors.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Pappas, PhD, Principal Investigator — Aspira Women's Health
Locations (10):
- United States (10):
  - New Horizons Clinical Trials, Chandler, Arizona
  - Velvet Clinical Research, Burbank, California
  - Reproductive Associates of Delaware (RAD), Newark, Delaware
  - Midtown OBGYN North, Columbus, Georgia
  - Cindy Basinski, MD, Forest Hill, Indiana
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Nezhat Surgery for Gynecology/Oncology, Valley Stream, New York
  - Seven Hills Clinical Research, Cincinnati, Ohio
  - May Grant, Lancaster, Pennsylvania
  - Womens Health Services of Central Virginia, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wykes CB, Clark TJ, Khan KS. Accuracy of laparoscopy in the diagnosis of endometriosis: a systematic quantitative review. BJOG. 2004 Nov;111(11):1204-12. doi: 10.1111/j.1471-0528.2004.00433.x. No abstract available. PMID 15521864
- [Background] Gupta D, Hull ML, Fraser I, Miller L, Bossuyt PM, Johnson N, Nisenblat V. Endometrial biomarkers for the non-invasive diagnosis of endometriosis. Cochrane Database Syst Rev. 2016 Apr 20;4(4):CD012165. doi: 10.1002/14651858.CD012165. PMID 27094925
- [Background] Revised American Society for Reproductive Medicine classification of endometriosis: 1996. Fertil Steril. 1997 May;67(5):817-21. doi: 10.1016/s0015-0282(97)81391-x. No abstract available. PMID 9130884